CLINICAL TRIAL: NCT02226276
Title: A Pilot Study of 64Cu-DOTA-Trastuzumab Positron Emission Tomography in Treatment of Advanced HER2 Positive Breast Cancer With the Antibody Drug Conjugate Ado-trastuzumab Emtansine
Brief Title: Copper Cu 64-DOTA-Trastuzumab PET in Predicting Response to Treatment With Ado-Trastuzumab Emtansine in Patients With Metastatic HER2 Positive Breast Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14099; NCI-2014-01812 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 14099 (Other: City of Hope Medical Center)
Record Dates: First submitted 2014-08-25; First posted 2014-08-27 (Estimated); Results first posted 2022-07-20 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Bone Metastases; HER2-positive Breast Cancer; Liver Metastases; Lung Metastases; Recurrent Breast Cancer; Soft Tissue Metastases; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; Trastuzumab; 64Cu-DOTA-trastuzumab; Ado-Trastuzumab Emtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (copper Cu 64-DOTA-trastuzumab PET) (Experimental): Patients undergo whole body fludeoxyglucose F 18 PET/CT. Patients then receive trastuzumab IV over 15 minutes immediately before receiving copper Cu 64-DOTA-trastuzumab IV and then undergo PET scans at 24 and 48 hours. Patients then receive ado-trastuzumab emtansine IV every 3 weeks until complete response or disease progression at the discretion of the treating oncologist. Patients undergo restaging by whole body fludeoxyglucose F 18 PET/CT every 6 weeks after initiation of treatment until disease progression.
  Interventions: Radiation: fludeoxyglucose F 18; Procedure: positron emission tomography; Procedure: computed tomography; Biological: trastuzumab; Radiation: copper Cu 64-DOTA-trastuzumab; Biological: ado-trastuzumab emtansine; Other: laboratory biomarker analysis

INTERVENTIONS:
Radiation: fludeoxyglucose F 18 — Undergo fludeoxyglucose F 18 PET/CT
  Other Names: 18FDG; FDG
Procedure: positron emission tomography — Undergo fludeoxyglucose F 18 PET/CT
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed
Procedure: computed tomography — Undergo fludeoxyglucose F 18 PET/CT
  Other Names: tomography, computed
Biological: trastuzumab — Given IV
  Other Names: anti-c-erB-2; Herceptin; MOAB HER2
Radiation: copper Cu 64-DOTA-trastuzumab — Given IV
  Other Names: 64Cu-DOTA-trastuzumab
Procedure: positron emission tomography — Undergo copper Cu-DOTA-trastuzumab PET
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed
Biological: ado-trastuzumab emtansine — Given IV
  Other Names: Kadcyla; T-DM1; trastuzumab-DM1; trastuzumab-MCC-DM1; trastuzumab-MCC-DM1 antibody-drug conjugate
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This pilot clinical trial studies how well copper Cu 64-tetra-azacyclododecanetetra-acetic acid (DOTA)-trastuzumab positron emission tomography (PET) works in predicting response to treatment with ado-trastuzumab emtansine in patients with human epidermal growth factor receptor 2 (HER2) positive breast cancer that has spread to other places in the body. Copper Cu 64-DOTA-trastuzumab is a chemotherapy drug (trastuzumab) attached to a radioactive substance. Diagnostic procedures using PET may allow scanners to take pictures of where the drug travels in the body and may help doctors identify which patients may benefit from treatment with ado-trastuzumab emtansine.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Correlate uptake of 64Cu-DOTA-trastuzumab (copper Cu 64-DOTA-trastuzumab) PET by individual tumors with subsequent tumor response to ado-trastuzumab emtansine as assessed by serial 18F-fludeoxyglucose (FDG) (fludeoxyglucose F 18)/PET-computed tomography (CT).

II. Compare tumor uptake of 64Cu-DOTA-trastuzumab PET between patients who do and patients who do not respond to ado-trastuzumab emtansine.

III. Obtain tumor tissue for subsequent assessment of the presence of putative molecular mechanisms of resistance (MMRs) to ado-trastuzumab emtansine. When funding becomes available, those samples will be used to explore the correlation between the presence of MMRs as assessed by histopathology and tumor response to ado-trastuzumab emtansine both in univariate analysis and in combination with tumor uptake of 64Cu-DOTA-trastuzumab as measured with PET/CT.

OUTLINE:

Patients undergo whole body fludeoxyglucose F 18 PET/CT. Patients then receive trastuzumab intravenously (IV) over 15 minutes immediately before receiving copper Cu 64-DOTA-trastuzumab IV and then undergo PET scans at 24 and 48 hours. Patients then receive ado-trastuzumab emtansine IV every 3 weeks until complete response or disease progression at the discretion of the treating oncologist. Patients undergo restaging by whole body fludeoxyglucose F 18 PET/CT every 6 weeks for 1 year after initiation of treatment until disease progression.

After completion of study treatment, patients are followed up for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be women who have histological confirmation of metastatic invasive breast cancer that has metastasized outside the region of the primary tumor and axilla; biopsy must be obtained prior to initiation of chemotherapy; it should be performed within 28 days prior to enrollment (patients with a biopsy of recurrent disease that is HER2-positive and have not received HER2-directed therapy since the biopsy can exceed the 28-day window up to 6 months); patients must have metastatic disease in lung, liver, soft-tissue or bone to qualify for the study (more than one site is permissible)
* At least 1 site of metastasis >= 20 mm in mean diameter must be identified
* The cancer must over express HER2 as determined by immunohistochemistry (IHC) and/or fluorescence in situ hybridization (FISH)
* Patients may not have received trastuzumab within 6 weeks of projected 64Cu-DOTA-trastuzumab/PET-CT
* Participants must have normal cardiac ejection fraction
* Ability to provide informed consent
* Patients that may need dose reduction to commence cycle 1 treatment
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Negative serum pregnancy test (female of childbearing potential only)
* Patients must have adequate cardiac function; left ventricular ejection fraction (LVEF) >= 50% as determined by multi gated acquisition (MUGA) scan or echocardiogram

Exclusion Criteria:

* Participants who have received trastuzumab within the prior 36 days
* Participants who are not considered candidates for ado-trastuzumab-emtansine
* No metastatic sites >= 20 mm
* Concurrent malignancy other than skin cancer - Inability to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-01-07; Primary Completion 2021-12-07 (Actual); Study Completion 2025-10-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Mortimer, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Diagnostic (Copper Cu 64-DOTA-trastuzumab PET): Patients undergo whole body fludeoxyglucose F 18 PET/CT. Patients then receive trastuzumab IV (45 mg) over 15 minutes immediately before receiving copper Cu 64-DOTA-trastuzumab IV (<15 mCi; protein dose 5 mg) and then undergo PET scans at 24 and 48 hours. Patients then receive ado-trastuzumab emtansine IV (3.6 mg/kg) every 3 weeks until complete response or disease progression at the discretion of the treating oncologist. Patients undergo restaging by whole body fludeoxyglucose F 18 PET/CT every 6 weeks after initiation of treatment until disease progression.
  fludeoxyglucose F 18: Undergo fludeoxyglucose F 18 PET/CT
  positron emission tomography: Undergo fludeoxyglucose F 18 PET/CT
  computed tomography: Undergo fludeoxyglucose F 18 PET/CT
  trastuzumab: Given IV
  copper Cu 64-DOTA-trastuzumab: Given IV
  positron emission tomography: Undergo copper Cu-DOTA-trastuzumab PET
  ado-trastuzumab emtansine: Given IV
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Diagnostic (Copper Cu 64-DOTA-trastuzumab PET)
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic (Copper Cu 64-DOTA-trastuzumab PET)
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 54 [46 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 6
  Asian | 2
  Hispanic | 1
  African American | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Relationship Between Average Tumor Uptake of Copper Cu 64-DOTA-trastuzumab as Measured by PET and Patient Best Response
Description: Relationship between patient best response to T-DM1 and measured tumor uptake of 64Cu-DOTA-trastuzumab employed a t-test with a 0.05 two-sided significance level comparing average uptake in responsive vs non-responsive patients. Tumor uptake measured as SUV defined as SUV = AC(tsc) Wb /[Dinj exp(-λ(tsc - tinj)] , where AC(tsc) is the activity concentration in the volume of interest (VOI, e. g., a tumor), Wb is the patient's body weight, Dinj is the activity injected at time tinj, and λ is the decay constant for the injected radioisotope. AC(tsc) is determined from the spatial density of counts acquired from the VOI. Tumor uptake was measured in terms of maximum voxel standardized uptake value, SUVmax. Response assessment adhered to Positron Emission Tomography (PET) Response Criteria in Solid Tumors (PERCIST 1.0).
Time Frame: Baseline
Measure: Median (Full Range); unit: SUVmax (g/mL)
Arm/Group | Diagnostic (Copper Cu 64-DOTA-trastuzumab PET)
Number analyzed (Participants) | 10
SUVmax (g/mL) | 3.1 [0.5 to 7]
Statistical Analysis 1: Comparison: Diagnostic (Copper Cu 64-DOTA-trastuzumab PET); Test type: Other; p < 0.05, t-test, 2 sided

2. Primary Outcome: Relationship Between Tumor Minimum Uptake of Copper Cu 64-DOTA-trastuzumab as Measured by PET and Patient Best Response
Description: Relationship between patient best response to T-DM1 and measured tumor uptake of 64Cu-DOTA-trastuzumab employed a t-test with a 0.05 two-sided significance level comparing minimum uptake in responsive vs non-responsive patients. Tumor uptake measured as SUV defined as SUV = AC(tsc) Wb /[Dinj exp(-λ(tsc - tinj)] , where AC(tsc) is the activity concentration in the volume of interest (VOI, e. g., a tumor), Wb is the patient's body weight, Dinj is the activity injected at time tinj, and λ is the decay constant for the injected radioisotope. AC(tsc) is determined from the spatial density of counts acquired from the VOI. Tumor uptake was measured in terms of minimum voxel standardized uptake value, SUVmin. Response assessment adhered to Positron Emission Tomography (PET) Response Criteria in Solid Tumors (PERCIST 1.0).
Time Frame: Up to 1 year
Measure: Median (Full Range); unit: SUVmin (g/mL)
Arm/Group | Diagnostic (Copper Cu 64-DOTA-trastuzumab PET)
Number analyzed (Participants) | 10
SUVmin (g/mL) | 5.1 [3 to 7]
Statistical Analysis 1: Comparison: Diagnostic (Copper Cu 64-DOTA-trastuzumab PET); Test type: Other; p < 0.01, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events occurred over a period of 3 years and 8 months.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Diagnostic (Copper Cu 64-DOTA-trastuzumab PET)
All-Cause Mortality (participants affected / at risk) | 2/10
Serious Adverse Events (participants affected / at risk) | 5/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diagnostic (Copper Cu 64-DOTA-trastuzumab PET) (N=10)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Confusion (Psychiatric disorders) | 1 (1)
Hallucinations (Psychiatric disorders) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diagnostic (Copper Cu 64-DOTA-trastuzumab PET) (N=10)
Anemia (Blood and lymphatic system disorders) | 9 (64)
bleeding from gums (Blood and lymphatic system disorders) | 1 (1)
bleeding from hard palate (Blood and lymphatic system disorders) | 1 (1)
bleeding from the hard palate (Blood and lymphatic system disorders) | 1 (3)
intermittent epistaxis - R nostril (Blood and lymphatic system disorders) | 1 (1)
intermittent nosebleed (Blood and lymphatic system disorders) | 1 (1)
lump in the R axilla (Blood and lymphatic system disorders) | 1 (4)
petechie (Blood and lymphatic system disorders) | 1 (2)
thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Aortic valve disease (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 5 (34)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
intermittent PVCs to auscultation (Cardiac disorders) | 1 (1)
intermittent tachycardia (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Cushingoid (Endocrine disorders) | 2 (11)
Hypothyroidism (Endocrine disorders) | 1 (42)
low cortisol level (Endocrine disorders) | 1 (1)
low cortisol level (under investigation with endocrinology) (Endocrine disorders) | 1 (2)
Blurred vision (Eye disorders) | 1 (6)
Decreased Peripheral Vision (Eye disorders) | 1 (3)
Decreased Peripheral dcreased (Eye disorders) | 1 (1)
Decreased Peripherla Vision (Eye disorders) | 1 (2)
Decreased Peropheral Vision (Eye disorders) | 1 (1)
Decreased peripherla vision (Eye disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Eyelid function disorder (Eye disorders) | 1 (2)
Photophobia (Eye disorders) | 1 (1)
Visual Symptoms (Eye disorders) | 1 (1)
Visual Symptoms (Eye disorders) | 1 (7)
Visual symptoms - only when she is tired (Eye disorders) | 1 (1)
decreased peripheral vision (Eye disorders) | 1 (10)
decreased peripheral vision after sugery (Eye disorders) | 1 (1)
decreased peripheral vision after surgery (Eye disorders) | 1 (5)
decreased peripheral vision after the 2/8 surgery (Eye disorders) | 1 (1)
decreased peripheral vision after the surger (Eye disorders) | 1 (1)
decreased peripheral vision after the surgery (Eye disorders) | 1 (8)
dicreased peripheral vision (Eye disorders) | 1 (1)
hyperropia (Eye disorders) | 1 (1)
intermittent blurry eye (Eye disorders) | 1 (1)
intermittent blurry eye (when reading for a long time) (Eye disorders) | 1 (1)
intermittent blurry eye when reads for long time (Eye disorders) | 1 (1)
photosensitivity (Eye disorders) | 1 (2)
shaking of eyes during C4 infusion (Eye disorders) | 1 (1)
shaking of eyes during trastuzumab emtansine infusion (Eye disorders) | 1 (1)
shaking of eyes during trastuzumab emtansive (Eye disorders) | 1 (1)
stye (Eye disorders) | 1 (1)
tired eyes - when reads for a long time (Eye disorders) | 1 (2)
tired eyes when reads for a long time (Eye disorders) | 1 (1)
visual symptoms (Eye disorders) | 1 (16)
visual symptoms (only when tired) (Eye disorders) | 1 (2)
visual symptoms - only when tired (Eye disorders) | 1 (1)
visual symptoms only when tired (Eye disorders) | 1 (1)
whipple in the left eye (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (11)
Bloating (Gastrointestinal disorders) | 2 (5)
Constipation (Gastrointestinal disorders) | 7 (32)
Diarrhea (Gastrointestinal disorders) | 4 (23)
Dry mouth (Gastrointestinal disorders) | 3 (19)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 4 (8)
Gastritis (Gastrointestinal disorders) | 1 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (3)
Heartburn (Gastrointestinal disorders) | 1 (8)
Mucositis oral (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 7 (75)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Tongue feels raw, Hurting (Gastrointestinal disorders) | 1 (1)
Tongue feels raw, hurting (Gastrointestinal disorders) | 1 (7)
Tounge feels raw, Hurting (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (17)
decreased appetite (Gastrointestinal disorders) | 1 (2)
epigastric discomfort (Gastrointestinal disorders) | 1 (2)
flactuating appetite after Keppra increased (Gastrointestinal disorders) | 1 (1)
glossitis (Gastrointestinal disorders) | 1 (1)
heartburn (Gastrointestinal disorders) | 1 (3)
increased appetite (Gastrointestinal disorders) | 1 (1)
increased thirst (Gastrointestinal disorders) | 1 (1)
indigestion (Gastrointestinal disorders) | 1 (2)
intermittent constipation (Gastrointestinal disorders) | 3 (11)
intermittent diarrhea (Gastrointestinal disorders) | 2 (4)
intermittent nausea (Gastrointestinal disorders) | 2 (15)
intermittent nausea - after Keppra increased (Gastrointestinal disorders) | 1 (1)
intermittent nausea after Keppra increased (Gastrointestinal disorders) | 1 (2)
intermittent rectal bleeding (Gastrointestinal disorders) | 1 (1)
intermittent vomiting (Gastrointestinal disorders) | 1 (1)
intermittent vomitting (Gastrointestinal disorders) | 1 (1)
low appetite (Gastrointestinal disorders) | 1 (1)
occasional blood in stool (Gastrointestinal disorders) | 1 (2)
occasional blood in stool while having hard stool (Gastrointestinal disorders) | 1 (1)
occasional constipation (Gastrointestinal disorders) | 1 (2)
plaque small white side of tongue (Gastrointestinal disorders) | 1 (2)
rectal bleeding (Gastrointestinal disorders) | 1 (1)
red, raw tongue (Gastrointestinal disorders) | 1 (1)
small white plaque L side of tongue (Gastrointestinal disorders) | 1 (1)
tenderness in mid-left abdomen w touch (Gastrointestinal disorders) | 1 (2)
tenderness in mid-left abdomen w/ touch (Gastrointestinal disorders) | 1 (1)
tongue feels raw, hurting (Gastrointestinal disorders) | 1 (2)
unable to eruct (Gastrointestinal disorders) | 1 (9)
Chills (General disorders) | 2 (2)
Edema limbs (General disorders) | 3 (6)
Fatigue (General disorders) | 10 (117)
Fever (General disorders) | 2 (5)
Flu like symptoms (General disorders) | 3 (4)
Localized edema (General disorders) | 1 (2)
Malaise (General disorders) | 1 (2)
Neck edema (General disorders) | 1 (2)
Non-cardiac chest pain (General disorders) | 2 (3)
Pain (General disorders) | 2 (2)
abscess (General disorders) | 1 (1)
low-grade temperature (General disorders) | 1 (1)
Rhinitis infective (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 1 (3)
Upper respiratory infection (Infections and infestations) | 2 (6)
Urinary tract infection (Infections and infestations) | 5 (8)
low grade temperature (Infections and infestations) | 1 (3)
oral thrush (Infections and infestations) | 1 (1)
shingles (Infections and infestations) | 1 (2)
suspected bacteremia (Infections and infestations) | 1 (1)
yeast infection (Infections and infestations) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 2 (9)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 5 (24)
Alkaline phosphatase increased (Investigations) | 7 (67)
Aspartate aminotransferase increased (Investigations) | 8 (71)
Creatinine increased (Investigations) | 2 (2)
Electrocardiogram QT corrected interval (Investigations) | 1 (1)
Hemoglobin increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 5 (19)
Neutrophil count decreased (Investigations) | 3 (13)
Platelet count decreased (Investigations) | 8 (95)
Weight gain (Investigations) | 2 (7)
White blood cell decreased (Investigations) | 4 (34)
Anorexia (Metabolism and nutrition disorders) | 7 (18)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (38)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (19)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (5)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (3)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 (19)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (6)
Hypokalemia (Metabolism and nutrition disorders) | 6 (23)
Hyponatremia (Metabolism and nutrition disorders) | 8 (35)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (2)
Obesity (Metabolism and nutrition disorders) | 1 (20)
occasional night sweats (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (2)
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 1 (28)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (8)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (6)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (5)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (11)
Joint range of motion decreased cervical (Musculoskeletal and connective tissue disorders) | 1 (1)
L ankle swelling and pain (Musculoskeletal and connective tissue disorders) | 1 (3)
L big toe bends in toward other toes (Musculoskeletal and connective tissue disorders) | 1 (3)
L big toe bends in towards other toes (Musculoskeletal and connective tissue disorders) | 1 (5)
L big toe bends toward other toes (Musculoskeletal and connective tissue disorders) | 1 (1)
L big toe bends towards other toes (Musculoskeletal and connective tissue disorders) | 1 (1)
L hand is curled inward (Musculoskeletal and connective tissue disorders) | 1 (1)
L shoulder and L middle finger joint pain (Musculoskeletal and connective tissue disorders) | 1 (4)
L shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1)
L sided limp (Musculoskeletal and connective tissue disorders) | 1 (2)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (10)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (8)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (9)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (13)
R elbow pain (Musculoskeletal and connective tissue disorders) | 1 (13)
R shoulder and arm pain (Musculoskeletal and connective tissue disorders) | 1 (2)
R shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (2)
R shoulder, arm pain (Musculoskeletal and connective tissue disorders) | 1 (1)
R shoulder/arm pain (Musculoskeletal and connective tissue disorders) | 1 (2)
arthritis R shoulder (Musculoskeletal and connective tissue disorders) | 1 (2)
avascular necrosis L humerus (Musculoskeletal and connective tissue disorders) | 1 (1)
bilateral elbow pain (Musculoskeletal and connective tissue disorders) | 1 (2)
bilateral shoulder and neck pain (Musculoskeletal and connective tissue disorders) | 1 (2)
bunionette (Musculoskeletal and connective tissue disorders) | 1 (1)
car accident injuries (Musculoskeletal and connective tissue disorders) | 1 (1)
car accident on 6/19/2018 (Musculoskeletal and connective tissue disorders) | 1 (1)
cramping (Musculoskeletal and connective tissue disorders) | 1 (1)
decreased mobility and pain in L arm (Musculoskeletal and connective tissue disorders) | 1 (1)
decreased mobility and pain in left arm/difficulty making fi (Musculoskeletal and connective tissue disorders) | 1 (1)
decreased mobility, pain left arm (Musculoskeletal and connective tissue disorders) | 1 (1)
decreased mobility, pain L arm (Musculoskeletal and connective tissue disorders) | 1 (1)
decreased mobility, pain L arm, difficulty making fist w L h (Musculoskeletal and connective tissue disorders) | 1 (1)
decreased mobility, pain L arm/difficulty making fist L hand (Musculoskeletal and connective tissue disorders) | 1 (2)
decreased mobility, pain in L arm (Musculoskeletal and connective tissue disorders) | 1 (1)
decreased mobility, pain left arm, difficulty making fist w (Musculoskeletal and connective tissue disorders) | 1 (1)
decreased mobility, pain left arm, difficulty making fist wi (Musculoskeletal and connective tissue disorders) | 1 (2)
decreased mobility/pain L arm, difficulty making fist L hand (Musculoskeletal and connective tissue disorders) | 1 (1)
decreased mobility/pain left arm, difficulty making fist wit (Musculoskeletal and connective tissue disorders) | 1 (1)
decreased mobility/pain left arm/difficulty making fist with (Musculoskeletal and connective tissue disorders) | 1 (1)
difficulty making fist with L arm (Musculoskeletal and connective tissue disorders) | 1 (1)
difficulty making fist with L hand (Musculoskeletal and connective tissue disorders) | 1 (4)
dupuytrens contracture status post surgery (Musculoskeletal and connective tissue disorders) | 1 (1)
intermittent L should pain - movement dependent (Musculoskeletal and connective tissue disorders) | 1 (1)
intermittent L shoulder pain - movement dependent (Musculoskeletal and connective tissue disorders) | 1 (6)
intermittent L shoulder pain movement dependent (Musculoskeletal and connective tissue disorders) | 1 (2)
intermittent bilateral rib pain (Musculoskeletal and connective tissue disorders) | 1 (3)
intermittent lower back pain (Musculoskeletal and connective tissue disorders) | 1 (6)
left shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (2)
mid-back pain (Musculoskeletal and connective tissue disorders) | 1 (5)
muscle cramps - both legs and back (Musculoskeletal and connective tissue disorders) | 1 (2)
neck stiffness (Musculoskeletal and connective tissue disorders) | 1 (4)
osteopenia (Musculoskeletal and connective tissue disorders) | 1 (23)
overall myalgia and body stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
pain and decreased mobility both arms (Musculoskeletal and connective tissue disorders) | 1 (1)
pain and decreased mobility in both arms (Musculoskeletal and connective tissue disorders) | 1 (1)
pain and swelling - back of L knee (Musculoskeletal and connective tissue disorders) | 1 (3)
pain in neck and shoulders (Musculoskeletal and connective tissue disorders) | 1 (1)
pain in the thighs (front of thighs and glutes) (Musculoskeletal and connective tissue disorders) | 1 (1)
pain in the thighs - front of thighs and glutes (Musculoskeletal and connective tissue disorders) | 1 (1)
right elbow pain (Musculoskeletal and connective tissue disorders) | 1 (1)
rotator cuff injury (Musculoskeletal and connective tissue disorders) | 1 (3)
rotator cuff injury R arm (Musculoskeletal and connective tissue disorders) | 1 (14)
shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1)
stiffness in knee and back (Musculoskeletal and connective tissue disorders) | 1 (1)
swollen area of R side of R foot (Musculoskeletal and connective tissue disorders) | 1 (1)
swollen area on R side of R foot (Musculoskeletal and connective tissue disorders) | 1 (2)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Ataxia (Nervous system disorders) | 1 (3)
Dizziness (Nervous system disorders) | 5 (14)
Dysgeusia (Nervous system disorders) | 2 (12)
Dysphasia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 4 (55)
L arm - pain of full abduction (Nervous system disorders) | 1 (2)
L arm - pain on full abduction (Nervous system disorders) | 1 (1)
L hand curled inward (Nervous system disorders) | 1 (13)
L side hemoplegia (Nervous system disorders) | 1 (1)
L side weak (as per getting up from squat, dragging) (Nervous system disorders) | 1 (2)
L sided hemiparesis (Nervous system disorders) | 1 (3)
L sided hemiplegia (Nervous system disorders) | 1 (14)
L sided hemoplegia (Nervous system disorders) | 1 (3)
L upper eyelid ptosis (Nervous system disorders) | 1 (2)
Lethargy (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (7)
Paresthesia (Nervous system disorders) | 2 (22)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 8 (62)
Recurrent laryngeal nerve palsy (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 2 (2)
intermittent dizziness w/ position change - preexisting as p (Nervous system disorders) | 1 (2)
intermittent dizziness w/ position change) (Nervous system disorders) | 1 (2)
intermittent headache (Nervous system disorders) | 2 (8)
intermittent headache (2 weeks after TX) (Nervous system disorders) | 1 (2)
intermittent headache (only scar pain when bends, lean over) (Nervous system disorders) | 1 (1)
intermittent headache (only scar pain, when bends, lean over (Nervous system disorders) | 1 (1)
intermittent sensitivity - feet - bottoms (Nervous system disorders) | 1 (1)
intermittent sensitivity - feet bottoms (Nervous system disorders) | 1 (1)
intermittent sensitivity feet botoms (Nervous system disorders) | 1 (1)
l sided hemiplegia (Nervous system disorders) | 1 (2)
left sided hemiplegia (Nervous system disorders) | 1 (3)
migraine (Nervous system disorders) | 1 (1)
pain at the base of the neck (Nervous system disorders) | 1 (1)
sensitivity - feet bottoms (Nervous system disorders) | 1 (1)
sensory neuropathy L arm (Nervous system disorders) | 1 (17)
sensory neuropathy left arm (Nervous system disorders) | 1 (3)
sensory neurophathy left arm (Nervous system disorders) | 1 (1)
vocal cord paralysis (Nervous system disorders) | 1 (3)
Agitation (Psychiatric disorders) | 2 (3)
Anxiety (Psychiatric disorders) | 3 (31)
Confusion (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (7)
Insomnia (Psychiatric disorders) | 2 (25)
anxiety re new brain lesions (Psychiatric disorders) | 1 (1)
emotional distress (Psychiatric disorders) | 1 (3)
Hematuria (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 2 (5)
UTI symptoms (dysuria, abdominal pain, changes in UA) (Renal and urinary disorders) | 1 (1)
UTI symptoms - dysuria, abdominal pain, changes in UA) (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
dysuria (Renal and urinary disorders) | 1 (2)
hot urine (Renal and urinary disorders) | 1 (1)
polyuria (Renal and urinary disorders) | 1 (2)
Irregular menstruation (Reproductive system and breast disorders) | 2 (6)
Vaginal hemorrhage (Reproductive system and breast disorders) | 2 (2)
candidiasis (Reproductive system and breast disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (29)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (15)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (44)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3 (9)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 (12)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (7)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
URI (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (7)
allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
allergic symptoms (Respiratory, thoracic and mediastinal disorders) | 1 (2)
allergies - patient reported (Respiratory, thoracic and mediastinal disorders) | 1 (1)
asthmatic bronchtis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
chest congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
cold symptoms (Respiratory, thoracic and mediastinal disorders) | 1 (1)
crackles in LLL (both insp and expiration) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
decreased O2 saturation (Respiratory, thoracic and mediastinal disorders) | 1 (8)
decreased oxygen saturation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
dry cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
dry cough (chronic as per patient), noted in the CRU (Respiratory, thoracic and mediastinal disorders) | 1 (1)
inspiratory crackles - left posterior lung base (Respiratory, thoracic and mediastinal disorders) | 1 (1)
intermittent chest discomofort (Respiratory, thoracic and mediastinal disorders) | 1 (1)
intermittent drippy nose following TX (Respiratory, thoracic and mediastinal disorders) | 1 (2)
intermittent drippy nose following treatment (Respiratory, thoracic and mediastinal disorders) | 1 (1)
intermittent dyspnea (only when activity and speech at the s (Respiratory, thoracic and mediastinal disorders) | 1 (3)
intermittent dyspnea only when activity and speech at the sa (Respiratory, thoracic and mediastinal disorders) | 1 (1)
occasional cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
occasional cough (provoked by food smell as per patient) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
occasional cough provoked by food smells as per patient (Respiratory, thoracic and mediastinal disorders) | 1 (1)
occasional sputum build up in the throat (Respiratory, thoracic and mediastinal disorders) | 1 (2)
occasional sputum build up in the troat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
possible small airway dysfunction (Respiratory, thoracic and mediastinal disorders) | 1 (6)
possible small airways dysfunction (Respiratory, thoracic and mediastinal disorders) | 1 (3)
productive cough w/ white or clear phlegm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
productive cough with white or clear phlegm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
rales and wheezes in LLL (Respiratory, thoracic and mediastinal disorders) | 1 (7)
rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
rhnorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
scattered wheezes R upper lobe (Respiratory, thoracic and mediastinal disorders) | 1 (1)
scattered wheezes in R upper lob (Respiratory, thoracic and mediastinal disorders) | 1 (2)
scattered wheezes in R upper lobe (Respiratory, thoracic and mediastinal disorders) | 1 (5)
scattered wheezes in the R upper lobe (Respiratory, thoracic and mediastinal disorders) | 1 (1)
small airway dysfunction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
sounds while sleeping (Respiratory, thoracic and mediastinal disorders) | 1 (3)
sputum build up in the throat (Respiratory, thoracic and mediastinal disorders) | 1 (3)
wheezing after excercise (Respiratory, thoracic and mediastinal disorders) | 1 (1)
wheezing after exercise (Respiratory, thoracic and mediastinal disorders) | 1 (1)
wheezing/cracking breath w/ expiration (Respiratory, thoracic and mediastinal disorders) | 1 (2)
worsening of L mid and lower lobe interst and ground glass o (Respiratory, thoracic and mediastinal disorders) | 1 (1)
worsening of L mid and lower lobe lung interst and ground gl (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (12)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (2)
Nail ridging (Skin and subcutaneous tissue disorders) | 1 (1)
Peeling of skin on feet (Skin and subcutaneous tissue disorders) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (34)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
capillary hemangioma (Skin and subcutaneous tissue disorders) | 1 (5)
erythema in response to RX therapy (Skin and subcutaneous tissue disorders) | 1 (1)
occasional pain in the incision area (Skin and subcutaneous tissue disorders) | 1 (1)
occasional soreness to the incision area (Skin and subcutaneous tissue disorders) | 1 (3)
occasional soreness to the incison area (Skin and subcutaneous tissue disorders) | 1 (1)
petechiae (Skin and subcutaneous tissue disorders) | 1 (3)
scabs and bruises on the back of L arm (Skin and subcutaneous tissue disorders) | 1 (2)
skin lesions from cupping (Skin and subcutaneous tissue disorders) | 1 (4)
skin lessions from cupping (Skin and subcutaneous tissue disorders) | 1 (1)
skin peeling at feet (Skin and subcutaneous tissue disorders) | 1 (1)
skin spot removed from the nose (Skin and subcutaneous tissue disorders) | 1 (1)
small raised bump on the R inner thigh (Skin and subcutaneous tissue disorders) | 1 (2)
sores on fingers (Skin and subcutaneous tissue disorders) | 1 (8)
weak nails (Skin and subcutaneous tissue disorders) | 1 (1)
menopausal like symptoms (Social circumstances) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 9 (119)
Hypotension (Vascular disorders) | 1 (11)
Lymphedema (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-18): https://cdn.clinicaltrials.gov/large-docs/76/NCT02226276/Prot_SAP_000.pdf